CLINICAL TRIAL: NCT05706662
Title: The DySLOH Study: Dynamic Scaffold Versus Lichtenstein Open Hernioplasty. A Comparative Outcome Assessment Between the Two Techniques.
Brief Title: Dynamic Scaffold Versus Lichtenstein Open Hernioplasty.
Acronym: DYSLOH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof. Antonino Agrusa, full professor of surgery, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DySLOH
Record Dates: First submitted 2023-01-21; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia repair; ProFlor technique; lichtenstein hernia repair
MeSH Terms: conditions — Hernia, Inguinal | interventions — Melanocyte-Stimulating Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ProFlor (Experimental): patients underwent to inguinal hernia repair with use of ProFlor dynamic scaffold
  Interventions: Procedure: inguinal hernia repair with mesh
- Lichtenstein (Active Comparator): patients underwent to Lichtenstein inguinal hernia repair
  Interventions: Procedure: inguinal hernia repair with mesh

INTERVENTIONS:
Procedure: inguinal hernia repair with mesh — inguinal hernia repair with mesh

SUMMARY:
Evaluating the outcomes of patients undergoing open anterior inguinal hernioplasty comparing two different techniques: Lichtenstein/plug and mesh and ProFlor. The outcomes of these two groups of patients, respectively the Lichtenstein inguinal hernia repair with static flat mesh and the defect obliteration with 3D dynamic scaffold Proflor, are compared in respect to defined variables along stages: intraoperative, early and long term postoperative.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients were individuals aged between 18 and 85 years old, competent to give consent, affected by clinically relevant primary inguinal hernia scheduled to undergo elective inguinal hernia repair and eligible for outpatient surgical procedure with local anesthesia.

Exclusion Criteria:

* Recurrent inguinal hernia
* Incarcerated inguinal hernia
* Hernia not in the inguinal area
* Signs of obvious local or systemic infection
* ASA score > 4
* Presenting with unstable angina or NYHA class of IV
* Pregnant
* Active drug user
* Immunosuppression, chemotherapy
* Chronic renal insufficiency
* Abdominal ascites
* Infection in area of the surgical field
* BMI >35

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
early postoperative complications | 30 days after surgery
  bleeding, hematoma and infections
patients clinical outcome | 24 months
  VAS score

SECONDARY OUTCOMES:
evaluation of quality of life during the postoperative period | 24 months
  Carolina Comfort Scale - CCS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No